CLINICAL TRIAL: NCT03683212
Title: Early and Comprehensive Care Bundle in Elderly for Acute Heart Failure: a Stepped Wedge Cluster Randomized Trial
Acronym: ELISABETH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: K170918J; 2018-A01139-46 (Other: ANSM)
Record Dates: First submitted 2018-07-09; First posted 2018-09-25 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Acute Heart Failure
Keywords: Emergency department; Elderly; Acute heart failure; Pulmonary edema
MeSH Terms: conditions — Emergencies; Pulmonary Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention period : early and comprehensive care bundle (Experimental)
  Interventions: Procedure: Early intensive care bundle
- acute heart failure standard therapy (No Intervention)

INTERVENTIONS:
Procedure: Early intensive care bundle — The care bundle comprises a list of items to follow and tick on a handover checklist within 4 hours of ED management:
  1. Treatment of the congestion: (international guidelines and recommendations)
  2. Treatment of precipitating factors
  3. NIV (non-invasive ventilation) if respiratory distress with hypercapnia and pH < 7.35 in absence of contra indication.
  4. Preventive LMWH (low molecular weight heparin) if no pre-existing anticoagulation therapy.
  Arms: Intervention period : early and comprehensive care bundle

SUMMARY:
This is a prospective multicentre (N=15), stepped-wedge randomized trial that aims to evaluate the benefit of a protocolised comprehensive care bundle for early management of acute heart failure in the ED.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is one of the most common diagnoses for elderly patients in the emergency department (ED), with an admission rate higher than 80% and 1-month mortality around 10%. There is scarce evidence of any clinical added value of a specific treatment to improve outcomes, and European guidelines for the management of AHF are based on moderate levels of evidence, due to the lack of randomized controlled trials. Recent reports suggest that the very early administration of full recommended therapy may decrease mortality. However, several studies highlighted that elderly patients often received suboptimal treatment: For example, less than a third of them received nitrates therapy while it is recommended. Furthermore, a recent preliminary study reported that only 50% of them are assessed for precipitating factors - although it has been reported that precipitating factors are independently associated with mortality.

The hypothesis of the Elisabeth Study s is that an early care bundle that comprises early and comprehensive management of symptoms, along with prompt detection and treatment of precipitating factors should improve AHF outcome in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and older admitted to the emergency department with a diagnosis of acute heart failure determined by the emergency physician, based on the presence of:

  * at least one of the following symptoms : acute, or worsening of dyspnea, orthopnea
  * one or more of the followings: pulmonary rales, peripheral edema, a chest radiograph or transthoracic echocardiography showing pulmonary vascular congestion signs, increased natriuretic peptides (BNP or NT-pro-BNP).
  * Patients affiliated to French social security ("AME excepted")
  * Written informed consent signed by the patient / the trustworthy person / family member / close relative, or inclusion in case of emergency and written informed consent will been signed by the patient (if need be by trustworthy person, family member or close relative) as soon as possible (article L1122-1-2 of the French Public Health Code)

Exclusion Criteria:

* Patients are excluded if they have any of the followings:

  * other obvious cause of acute illness (severe sepsis, ST elevation Myocardial infarction)
  * systolic blood pressure less than 100 mmHg
  * severe mitral or aortic stenosis, or severe aortic regurgitation
  * known chronic kidney injury on dialysis
  * shock from any cause
  * Time from ED entrance to inclusion > 6h
* Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 503 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Number of days alive and out of hospital | 30 days
  Number of days alive and out of hospital

SECONDARY OUTCOMES:
To evaluate the effect of AHF management on the 30-day cardiovascular death | 30 days
  cardiovascular death
To evaluate the effect of AHF management on the 30-day all causes death | 30 days
  all causes death
To evaluate the effect of AHF management on the hospital readmission at 30 days | 30 days
  hospital readmission
To evaluate the effect of AHF management on the length of stay in hospital | 30 days
  length of stay in hospital
To evaluate the effect of AHF management on changes of more than 2 fold in creatinine level from randomization to day 30 or to discharge whichever comes first | 30 days
  creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freund Y, Cachanado M, Delannoy Q, Laribi S, Yordanov Y, Gorlicki J, Chouihed T, Feral-Pierssens AL, Truchot J, Desmettre T, Occelli C, Bobbia X, Khellaf M, Ganansia O, Bokobza J, Balen F, Beaune S, Bloom B, Simon T, Mebazaa A. Effect of an Emergency Department Care Bundle on 30-Day Hospital Discharge and Survival Among Elderly Patients With Acute Heart Failure: The ELISABETH Randomized Clinical Trial. JAMA. 2020 Nov 17;324(19):1948-1956. doi: 10.1001/jama.2020.19378. PMID 33201202
- [Derived] Freund Y, Gorlicki J, Cachanado M, Salhi S, Lemaitre V, Simon T, Mebazaa A. Early and comprehensive care bundle in the elderly for acute heart failure in the emergency department: study protocol of the ELISABETH stepped-wedge cluster randomized trial. Trials. 2019 Jan 31;20(1):95. doi: 10.1186/s13063-019-3188-8. PMID 30704508